CLINICAL TRIAL: NCT05068661
Title: A Randomized Controlled Trial of Combined Spinal Epidural Versus Dural Puncture Epidural Techniques for Labor Analgesia
Brief Title: Comparing Effectiveness of CSE Versus DPE for Labor Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00108996
Record Dates: First submitted 2021-09-13; First posted 2021-10-06 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Labor Pain
Keywords: labor analgesia; neuraxial technique; combined spinal epidural; dural puncture epidural
MeSH Terms: conditions — Labor Pain | interventions — Ropivacaine; Fentanyl; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Spinal Epidural (Active Comparator): 10 mcg of preservative-free fentanyl and 2 mg of preservative-free isobaric 0.25% bupivacaine will be administered into the intrathecal space to initiate analgesia. Labor analgesia will be maintained by programmed intermittent bolus with patient-controlled epidural analgesia (PCEA) as per standard of care.
  Interventions: Drug: Ropivacaine 0.1% Injectable Solution; Drug: Bupivacaine 0.25% Injectable Solution
- Dural Puncture Epidural (Active Comparator): A 25-G Whitacre needle will be used to puncture the dura. An initiation dose of 20 mL of ropivacaine 0.1% with fentanyl (2 mcg/mL) will be administered. Labor analgesia will be maintained by programmed intermittent bolus with patient-controlled epidural analgesia (PCEA) as per standard of care.
  Interventions: Drug: Ropivacaine 0.1% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.1% Injectable Solution — DPE
  Other Names: Fentanyl
Drug: Bupivacaine 0.25% Injectable Solution — CSE
  Other Names: Ropivacaine 0.1% Injectable Solution; Fentanyl
  Arms: Combined Spinal Epidural

SUMMARY:
The primary purpose of this study is to determine if there are differences in block quality between the CSE and DPE techniques for labor analgesia in parturients in active labor. We hypothesize that when compared to the CSE technique, the DPE technique will significantly improve block quality in this population and require fewer "top-ups" and catheter replacements.

DETAILED DESCRIPTION:
This will be a prospective, double-blinded, randomized trial.

Subject identification and recruitment:

Women admitted to the Duke Birthing Center for spontaneous or induced labor will be screened. After usual consultation with the anesthesia team is completed and consent for anesthesia services are obtained, eligible patients will be approached to by a member of the study team. As indicated below, we will plan to enroll up to 120 patients to have 100 patients with complete data (50 for the CSE group and 50 for the DPE group).

Assignment of Study Cohorts:

Study participants will be randomized by computer-generated sequence to CSE or DPE arms, stratified by parity (nulliparous versus multiparous). After the consented and enrolled participant requests labor epidural, a study member will give the anesthesia provider a sealed envelope with study assignment for either standard CSE or DPE technique.

Epidural technique:

Once the patient requests labor analgesia, the usual standard of care for epidural placement will be initiated. The patient will receive 500-1000 mL fluid preload. Vitals will be monitored by the labor nurse, including continuous pulse oximetry, non-invasive blood-pressure monitoring, and external tocodynamometry. Anesthesia time-out will be performed by the anesthesia provider with participation from the nurse and the patient.

All patients will receive a neuraxial technique in the sitting position at L3/4 or L4/5 using loss of resistance to saline. In both the CSE and DPE groups, a 25-G Whitacre needle will be used to puncture the dura. In the CSE group, 10 mcg of preservative-free fentanyl and 2 mg of preservative-free isobaric 0.25% bupivacaine will be administered into the intrathecal space. In both groups, the epidural catheter will be threaded 5 cm into the epidural space. In the DPE group, an initiation dose of 20 mL of ropivacaine 0.1% with fentanyl (2 mcg/mL) over 6 minutes. This would not be administered in the CSE group. Labor analgesia will be maintained by programmed intermittent bolus with 8 mL of the same solution every 45 minutes starting 30 minutes after the initial dose. Patients will have patient-controlled epidural analgesia (PCEA) available with an 10 mL dose per demand, every 10 minutes, for a maximum dose of 50 mL for every hour.

Data Collection:

After the block is placed, a blinded provider will enter the room to collect data. Data will be collected every 3 minutes for the first 30 minutes or until pain score is 1 or 0 with uterine contractions. Subsequent assessments will be every 2 hours until delivery.

Management of breakthrough pain will be standardized.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45, singleton, vertex fetuses at 37-41 weeks' gestation, nulliparous and multiparous women, cervical dilation of 2-7cm, pain score > 4, and English-speaking ability

Exclusion Criteria:

* Women with major cardiac disease, chronic pain, chronic opioid use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women who have a singleton pregancy at 37-41 weeks' gestation
Enrollment: 101 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf S Habib, MD, Principal Investigator — Duke University Hospital
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
Started | 49 | 52
Completed | 48 | 52
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (5) | 32 (4) | 32 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 41 | 47 | 88
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 12 | 21
  White | 29 | 30 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 52 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Presence of Any of the Five Block Quality Components (or More Than One)
Description: The primary outcome of this study is block quality which will be defined by a composite of five components (1) asymmetric block after 30 minutes of initiation, (2) top-up interventions, (3) catheter adjustments (4) failed catheter requiring replacement, and (5) failed epidural requiring general anesthesia or replacement neuraxial anesthesia for cesarean section. The presence of any of the components (or more than one) indicates that the outcome occurred.
Time Frame: From placement of epidural to delivery of baby, up to 32 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
Number analyzed (Participants) | 48 | 52
Participants | 16 | 13
Statistical Analysis 1: Comparison: Combined Spinal Epidural vs Dural Puncture Epidural; Test type: Superiority; p = 0.486, Chi-squared; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.40 to 1.39]

2. Secondary Outcome: Maternal Adverse Events
Description: This will include instances such as: hypotension defined as 20% drop in blood pressure from admission blood pressure, fetal bradycardia, PDPH
Time Frame: From placement of epidural to delivery, up to 32 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
Number analyzed (Participants) | 48 | 52
Participants | 40 | 37
Statistical Analysis 1: Comparison: Combined Spinal Epidural vs Dural Puncture Epidural; Test type: Superiority; p = 0.148, Chi-squared — This is adjusted P value for hypotension; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.69 to 1.06]

3. Secondary Outcome: Number of Participants With Motor Block as Measured by the Modified Bromage Score
Description: Motor block is defined as a Bromage score of 1 to 4 on a scale of 1 to 5. 1 = unable flex feet or knees, 2 = able to flex feet only, 3 = able to flex knees, 4 = detectable weakness in hip flexion, 5 = no weakness in hip flexion.
Time Frame: From placement of epidural to delivery, up to 32 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
Number analyzed (Participants) | 48 | 52
Participants | 13 | 10
Statistical Analysis 1: Comparison: Combined Spinal Epidural vs Dural Puncture Epidural; Test type: Superiority; p > 0.999, Chi-squared — This is adjusted P value; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.98 to 1.10]

4. Secondary Outcome: Duration of the Second Stage of Labor
Description: Time from initiation of pushing to delivery of baby will be recorded
Time Frame: From start of second stage of labor to delivery, up to 6 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
Number analyzed (Participants) | 48 | 52
minutes | 23 [10 to 57] | 47 [20 to 97]
Statistical Analysis 1: Comparison: Combined Spinal Epidural vs Dural Puncture Epidural; Test type: Superiority; p = 0.128, Regression, Linear — Adjusted P value; Mean Ratio = 1.90, 95% CI 2-sided [1.14 to 3.18]

5. Secondary Outcome: Total Labor Epidural Time
Description: Time from placement of epidural to delivery will be recorded in anesthetic record
Time Frame: From placement of epidural to delivery, up to 32 hours
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
Number analyzed (Participants) | 48 | 52
Minutes | 443 [304 to 738] | 534 [292 to 747]
Statistical Analysis 1: Comparison: Combined Spinal Epidural vs Dural Puncture Epidural; Test type: Superiority; p > 0.999, Regression, Linear — Adjusted P value; Mean Ratio = 1.04, 95% CI 2-sided [0.80 to 1.35]

6. Secondary Outcome: Total Anesthetic Dose Required
Description: Total volume of local anesthetic will be recorded.
Time Frame: From placement of epidural to delivery, up to 32 hours
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
Number analyzed (Participants) | 48 | 52
mL | 108 [81 to 143] | 108 [65 to 162]
Statistical Analysis 1: Comparison: Combined Spinal Epidural vs Dural Puncture Epidural; Test type: Superiority; p > 0.999, Regression, Linear — Adjusted P value; Mean Ratio = 0.97, 95% CI 2-sided [0.93 to 1.30]

7. Secondary Outcome: Number of Participants Who Self-administered PCEA (Patient-controlled Epidural Analgesia) Boluses
Time Frame: From placement of epidural to delivery, up to 32 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
Number analyzed (Participants) | 48 | 52
Participants | 40 | 41
Statistical Analysis 1: Comparison: Combined Spinal Epidural vs Dural Puncture Epidural; Test type: Superiority; p > 0.999, Chi-squared — Adjusted P value; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.52 to 1.25]

8. Secondary Outcome: Mode of Delivery
Description: Spontaneous and assisted deliveries will be recorded
Time Frame: Through completion of the study, up to 32 hours from epidural placement
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
Number analyzed (Participants) | 48 | 52
Participants
  Spontaneous Vaginal Delivery | 32 | 33
  Forceps Assisted Delivery | 2 | 1
  Vacuum Assisted Delivery | 1 | 0
  Cesarean Delivery | 13 | 18
Statistical Analysis 1: Comparison: Combined Spinal Epidural vs Dural Puncture Epidural; Test type: Superiority; p > 0.999, Chi-squared — Adjusted P value; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.58 to 1.24]

9. Secondary Outcome: Postpartum: Satisfaction With Analgesia Overall
Description: Patient satisfaction scores will be recorded from scale of 0 to 10, with 10 being the highest level of satisfaction
Time Frame: From placement of epidural to delivery, up to 32 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale (0-10)
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
Number analyzed (Participants) | 48 | 52
score on a scale (0-10) | 10 [8 to 10] | 10 [8 to 10]
Statistical Analysis 1: Comparison: Combined Spinal Epidural vs Dural Puncture Epidural; Test type: Superiority; p > 0.999, Regression, Linear — Adjusted P value; Mean Ratio = 1.03, 95% CI 2-sided [0.86 to 1.22]

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Combined Spinal Epidural | Dural Puncture Epidural
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/52
Other Adverse Events (participants affected / at risk) | 40/48 | 37/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Spinal Epidural (N=48) | Dural Puncture Epidural (N=52)
Hypotension (Vascular disorders) | 8 (8) | 11 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 38 (38) | 30 (30)
Nausea (Gastrointestinal disorders) | 13 (13) | 16 (16)
Postdural Puncture Headache (Nervous system disorders) | 1 (1) | 0 (0)
Fetal Heart Rate decelerations (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT05068661/Prot_SAP_000.pdf